CLINICAL TRIAL: NCT05032157
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study of Remibrutinib (LOU064) to Investigate the Efficacy, Safety and Tolerability for 52 Weeks in Adult Chronic Spontaneous Urticaria (CSU) Patients Inadequately Controlled by H1-antihistamines
Brief Title: A Phase 3 Study of Efficacy and Safety of Remibrutinib in the Treatment of CSU in Adults Inadequately Controlled by H1-antihistamines
Acronym: REMIX-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064A2302; 2021-000424-35 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-09-02 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Bruton Tyrosine Kinase (BTK) inhibitor; Chronic Spontaneous Urticaria (CSU); Urticaria Activity Score (UAS); Weekly Urticaria Activity Score (UAS7); Hives Severity Score (HSS); Weekly Hives Severity Score (HSS7); Itch Severity Score (ISS); Weekly Itch Severity Score (ISS7); Angioedema Activity Score (AAS); Weekly Angioedema Activity Score (AAS7); Dermatology Life Quality Index (DLQI)
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LOU064 25mg b.i.d. (Experimental): LOU064A (blinded) taken orally b.i.d. for 24 weeks, followed by LOU064 (open- label) taken orally b.i.d. for 28 weeks. Randomised in 2:1 ratio (active vs placebo)
  Interventions: Drug: LOU064 (blinded); Drug: LOU064 (open-label)
- Placebo (Placebo Comparator): LOU064A placebo (blinded) taken orally for 24 weeks, followed by LOU064 (open-label) taken orally b.i.d. for 28 weeks. Randomised in 2:1 ratio (active vs placebo)
  Interventions: Drug: Placebo; Drug: LOU064 (open-label)

INTERVENTIONS:
Drug: LOU064 (blinded) — LOU064 (blinded) active treatment
  Other Names: remibrutinib
  Arms: LOU064 25mg b.i.d.
Drug: Placebo — Placebo
  Arms: Placebo
Drug: LOU064 (open-label) — LOU064 (open-label) active treatment
  Other Names: remibrutinib

SUMMARY:
The purpose of this study was to establish the efficacy, safety, and tolerability of Remibrutinib 25 mg b.i.d. in adult patients suffering from chronic spontaneous urticaria (CSU) inadequately controlled by second generation H1-antihistamines (H1-AHs) in comparison to placebo.

DETAILED DESCRIPTION:
The study consisted of four periods, the total study duration was up to 60 weeks: Screening period of up to 4 weeks, Double-blind placebo-controlled treatment period of 24 weeks, Open-label treatment period with Remibrutinib period of 28 weeks, and treatment free follow-up period of 4 weeks.

The design of this study was a replicate of another Phase III study, CLOU046A2301 (NCT05030311).

The study population consisted of female and male adult patients with CSU inadequately controlled by second generation H1-AHs at least at a locally label approved dose. All patients were on a stable, locally label approved dose of a second generation H1 AH (background therapy) throughout the entire study (starting a minimum of 7 days prior to randomization until the end of the study). To treat unbearable symptoms of CSU, patients were allowed to use another second generation H1-AH on an as-needed basis (rescue therapy). Eligible patients were randomly assigned to the treatment arms in a 2:1 ratio to remibrutinib or placebo arm (300 in the remibrutinib arm and 150 in placebo arm) and stratified based on prior exposure to anti-IgE biologics for CSU and geographic region.

An extension Phase IIIb study, CLOU064A2303B (NCT05513001), was initiated to allow CLOU064A2302 eligible patients to roll over after completion of the open-label treatment period.

There were two distinct testing strategies (scenario 1 with Weekly Urticaria Activity Score (UAS7) as the primary efficacy endpoint and scenario 2 with Weekly Itch Severity Score (ISS7) and Weekly Hives Severity Score (HSS7) as the co-primary efficacy endpoints) based on two primary objective scenarios related to regional regulatory precedent and Health Authorities' feedback.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male and female adult participants >= 18 years of age at the time of screening.
* CSU duration for >= 6 months prior to screening (defined as the onset of CSU determined by the investigator based on all available supporting documentation).
* Diagnosis of CSU inadequately controlled by second generation H1-antihistamines at the time of randomization defined as:

  * The presence of itch and hives for >= 6 consecutive weeks prior to screening despite the use of second generation H1-antihistamines during this time period
  * UAS7 score (range 0-42) >= 16, ISS7 score (range 0-21) >= 6 and HSS7 score (range 0-21) >= 6 during the 7 days prior to randomization (Day 1)
* Documentation of hives within three months before randomization (either at screening and/or at randomization; or documented in the participants medical history).
* Willing and able to complete an Urticaria Patient Daily Diary (UPDD) for the duration of the study and adhere to the study protocol.
* Participants must not have had more than one missing UPDD entry (either morning or evening) in the 7 days prior to randomization (Day 1).

Key Exclusion Criteria:

* Participants having a clearly defined predominant or sole trigger of their chronic urticaria (CU) (chronic inducible urticaria (CINDU)) including urticaria factitia (symptomatic dermographism), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
* Other diseases with symptoms of urticaria or angioedema, including but not limited to urticaria vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary urticaria, or drug-induced urticaria
* Any other skin disease associated with chronic itching that might influence in the investigator's opinion the study evaluations and results, e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or psoriasis
* Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, New York heart association (NYHA) Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 12 months prior to Visit 1), neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant
* Significant bleeding risk or coagulation disorders
* History of gastrointestinal bleeding, e.g. in association with use of nonsteroidal anti-inflammatory drugs (NSAID), that was clinically relevant (e.g. requiring hospitalization or blood transfusion)
* Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel. The use of dual anti-platelet therapy (e.g. acetylsalicylic acid + clopidogrel) is prohibited.
* Requirement for anticoagulant medication (for example, warfarin or Novel Oral Anti-Coagulants (NOAC))
* History or current hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure or Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) levels of more than 1.5 x upper limit of normal (ULN) or International Normalized Ratio (INR) of more than 1.5 at screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (111):
- United States (30):
  - Cahaba Derm and skin hlth ctr 27, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Little Rock Allergy and Asthma Clnc, Little Rock, Arkansas
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - UCONN Health Dermatology, Farmington, Connecticut
  - Miami Dade Medical Research, Miami, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Riverchase Dermatology, Pembroke Pines, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - AeroAllergy Research Laboratories of Savannah Inc, Savannah, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Northshore University Health System, Glenview, Illinois
  - Asthma and Allergy Center of Chicago S C, River Forest, Illinois
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - John Hopkins University, Baltimore, Maryland
  - Chesapeake Clinical Research, White Marsh, Maryland
  - Revival Research Institute, Troy, Michigan
  - Montana Medical Research, Missoula, Montana
  - Allergy Asthma Assoc Monmouth, Little Silver, New Jersey
  - Peters Medical Research, High Point, North Carolina
  - CR Services Acquisition US, Dublin, Ohio
  - Ohio Clinical Research Associates, Mayfield Heights, Ohio
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research LLS, North Charleston, South Carolina
  - STAAMP Research LLC, San Antonio, Texas
  - Intermountain Clinical Research, Salt Lake City, Utah
  - Seattle Allergy and Asthma Rsch, Seattle, Washington
  - Allergy Asthma and amp Sinus Ctr S C, Greenfield, Wisconsin
- Novartis Investigative Site, Linz, Upper Austria, Austria
- Novartis Investigative Site, São Bernardo do Campo, São Paulo, Brazil
- Canada (8):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Fredericton, New Brunswick
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Verdun, Quebec
- China (12):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Guangdong, Guangzhou
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Yiwu, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Denmark (2):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hellerup
- Germany (16):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bramsche
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Merzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- India (9):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Surat
- Malaysia (5):
  - Novartis Investigative Site, Muar town, Johor
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Pulau Pinang
  - Novartis Investigative Site, Wilayah Persekutuan
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Slovakia (4):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Topoľčany
- South Africa (3):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Cape Town, Western Province
  - Novartis Investigative Site, Cape Town
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taoyuan District
- Thailand (4):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (3):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Oxford
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Metz M, Gimenez-Arnau A, Hide M, Lebwohl M, Mosnaim G, Saini S, Sussman G, Szalewski R, Haemmerle S, Lheritier K, Martzloff ED, Seko N, Wang P, Zharkov A, Maurer M; REMIX-1 and REMIX-2 Investigators; REMIX-1 Investigators; REMIX-2 Investigators. Remibrutinib in Chronic Spontaneous Urticaria. N Engl J Med. 2025 Mar 6;392(10):984-994. doi: 10.1056/NEJMoa2408792. PMID 40043237
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted globally across 18 countries: Austria (1 center), Brazil (1 center), Canada (8 centers), China (16 centers), Denmark (2 centers), Germany (18 centers), India (10 centers), Malaysia (5 centers), Poland (5 centers), Russia (5 centers), Slovakia (4 centers), South Africa (3 centers), Switzerland (3 centers), Taiwan (2 centers), Thailand (4 centers), United Kingdom (3 centers), USA (30 centers), and Vietnam (2 centers).
Pre-assignment Details: Participants underwent a screening period of up to 4 weeks.
Groups:
- LOU064 25 mg b.i.d.: Patients initially randomized to Remibrutinib during the Double-blind treatment period and continued Remibrutinib during the Open-label treatment period (Up to Week 52)
- Placebo: Patients initially randomized to Placebo during the Double-Blind treatment period (Up to Week 24)
Period: Overall Study
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Started (All randomized patients, regardless of whether or not they received a dose of study drug.) | 300 | 155
Full Analysis Set (FAS) (All patients to whom study treatment was assigned by randomization. Mis-randomized patients were excluded from FAS.) | 297 | 153
Safety Set (SAF) (All patients who received at least one dose of study treatment, whether or not randomized.) | 297 | 153
Completed | 230 | 111
Not Completed | 70 | 44
Not completed — Adverse Event | 12 | 7
Not completed — Pregnancy | 0 | 2
Not completed — Unsatisfactory therapeutic effect | 4 | 7
Not completed — Protocol Deviation | 8 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 7 | 2
Not completed — Patient Decision | 38 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOU064 25 mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 300 | 155 | 455
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (14.52) | 41.3 (14.58) | 41.7 (14.53)
Age, Customized [Count of Participants; unit: Participants]
  >= 18 and < 65 years | 276 | 144 | 420
  >= 65 and < 85 years | 24 | 11 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 100 | 297
  Male | 103 | 55 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 130 | 72 | 202
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 159 | 79 | 238
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 12 (Scenario 1 With UAS7 as Primary Efficacy Endpoint)
Description: The Weekly Urticaria Activity Score (UAS7) is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42 (highest urticaria severity), and a minimum possible score of 0.
  This endpoint is a secondary endpoint for testing strategy Scenario 2 with Weekly Itch Severity Score (ISS7) and Weekly Hives Severity Score (HSS7) as co-primary efficacy endpoints).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Unit on a scale | -19.41 (0.702) | -11.73 (0.948)
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; UAS7 at Week 12 (Scenario 1 with UAS7 as primary efficacy endpoint); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -7.68, 95% CI 2-sided [-9.91 to -5.46], Standard Error of Mean 1.136 — MMRM adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics, week, baseline score and both interaction of treatment by week and interaction of baseline score by week

2. Primary Outcome: Mean Change From Baseline in Weekly Itch Severity Score (ISS7) at Week 12 (Scenario 2 With ISS7 and HSS7 as Co-primary Efficacy Endpoints)
Description: The severity of the itch was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (severe). A weekly score (ISS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest itch severity).
  This endpoint is a secondary endpoint for testing strategy Scenario 1 with Weekly Urticaria Activity Score (UAS7) as the primary efficacy endpoint).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Unit on a scale | -8.95 (0.335) | -5.72 (0.454)
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; ISS7 at Week 12 (Scenario 2 with ISS7 and HSS7 as co-primary efficacy endpoints); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.23, 95% CI 2-sided [-4.29 to -2.16], Standard Error of Mean 0.545 — MMRM adjusting for treatment arm, geographical region, prior exposure to anti- IgE, biologics, week, baseline score, and both interaction of treatment by week and interaction of baseline score by week

3. Primary Outcome: Mean Change From Baseline in Weekly Hives Severity Score (HSS7) at Week 12 (Scenario 2 With ISS7 and HSS7 as Co-primary Efficacy Endpoints)
Description: The hives (wheals) severity score, defined by number of hives, was recorded by the participant twice daily in their electronic Diary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest hives activity).
  This endpoint is a secondary endpoint for testing strategy Scenario 1 with Weekly Urticaria Activity Score (UAS7) as the primary efficacy endpoint).
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Unit on a scale | -10.47 (0.394) | -6.00 (0.531)
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; HSS7 at Week 12 (Scenario 2 with ISS7 and HSS7 as co-primary efficacy endpoints); Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.47, 95% CI 2-sided [-5.71 to -3.23], Standard Error of Mean 0.634 — MMRM adjusting for treatment arm, geographical region, prior exposure to anti- IgE biologics, week, baseline score and both interaction of treatment by week and interaction of baseline score by week

4. Secondary Outcome: Number of Participants Who Achieved Disease Activity Control (UAS7 =< 6) at Week 12
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Participants | 139 | 30
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Disease activity control (UAS7 =< 6) at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.84, 95% CI 2-sided [2.39 to 6.18] — Logistic regression adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics, and baseline UAS7 score

5. Secondary Outcome: Number of Participants Who Achieved Complete Absence of Hives and Itch (UAS7 = 0) at Week 12
Description: The proportion of patients achieving complete absence of hives and itch (UAS7 = 0) at Week 12 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Participants | 83 | 10
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Complete absence of hives and itch (UAS7 = 0) at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.78, 95% CI 2-sided [2.83 to 11.78] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Number of Participants Who Achieved Early Onset of Disease Activity Control (UAS7 =< 6) at Week 2
Description: The percentage of patients achieving disease activity control (UAS7 =< 6) at Week 2 was assessed to evaluate the efficacy of Remibrutinib in Chronic Spontaneous Urticaria (CSU) patients. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Week 2
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Participants | 89 | 9
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Early onset of disease activity control (UAS7 =< 6) at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.92, 95% CI 2-sided [3.72 to 16.85] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Number of Participants Who Achieved Dermatology Life Quality Index (DLQI) = 0-1 at Week 12
Description: The Dermatology Life Quality Index (DLQI) is a 10-item (grouped in 6 domains) dermatology-specific quality of life (QoL) measure. Participants are rating their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease-related QoL). Domain scores are calculated for: Symptoms and Feelings (0-6), Daily Activities (0-6), Leisure (0-6), Work and School (0-3), Personal Relationships (0-6), Treatment (0-3). The overall DLQI score range was split into score bands and validated in terms of their meaning/relevance to patients overall DLQI = 0-1 means no effect on patient's life.
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Participants | 106 | 28
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Dermatology Life Quality Index (DLQI) = 0-1 at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.75, 95% CI 2-sided [1.65 to 4.58] — Logistic regression adjusting for treatment arm, geographical region, prior exposure to anti-IgE biologics and baseline DLQI score

8. Secondary Outcome: Mean Cumulative Number of Weeks With Disease Activity Control (UAS7 =< 6) up to Week 12
Description: Maintaining disease activity control was assessed as cumulative number of weeks with an UAS7 =< 6 response between baseline and Week 12. The UAS7 is the sum of the Weekly Hives Severity Score (HSS7) and the Weekly Itch Severity Score (ISS7). The possible range of the UAS7 score is 0 - 42 (highest hives and itch severity).
Time Frame: Up to Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Weeks | 4.50 (0.464) | 1.38 (0.216)
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Disease activity control (UAS7 =< 6) up to Week 12; Test type: Superiority; p < 0.001, Regression, Linear; Rate ratio = 3.26, 95% CI 2-sided [2.26 to 4.71] — Negative binomial regression with log link includes treatment arm as fixed effect, geographical region, prior exposure to anti-IgE biologics as covariates. A rate ratio >1 favors LOU064 25 mg b.i.d

9. Secondary Outcome: Mean Cumulative Number of Angioedema Occurrence-free Weeks (AAS7 = 0 Response) up to Week 12
Description: Angioedema occurrence was recorded once daily in the evening in the electronic Diary by the participant. Reporting the occurrence of angioedema was used as opening question for the assessment of the Angioedema Activity Score (AAS). The AAS consists of 5 questions with 4 answer options (scored 0-3) for each item, with a minimum score of 0 and a maximum score of 15 per day. The AAS score over 7 days (AAS7) ranges from 0 (no angioedema episodes) to 105 (highest angioedema severity).
Time Frame: Up to Week 12
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | LOU064 25 mg b.i.d. | Placebo
Number analyzed (Participants) | 297 | 153
Weeks | 8.81 (0.308) | 6.68 (0.343)
Statistical Analysis 1: Comparison: LOU064 25 mg b.i.d. vs Placebo; Angioedema occurrence-free weeks (AAS7 = 0 response) up to Week 12; Test type: Superiority; p < 0.001, Regression, Linear; Rate ratio = 1.32, 95% CI 2-sided [1.17 to 1.49] — Negative binomial regression with log link included treatment arm as fixed effect, geographical region, prior exposure to anti-IgE biologics, baseline AAS7 = 0 response as covariates. A rate ratio > 1 favors LOU064 25 mg b.i.d

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Treatment emergent Adverse Event (TEAEs) in this study are events that started after the first dose of study treatment and until 28 days after the last dose of study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 28 days after the last study treatment.
Time Frame: Baseline up to 28 days after last dose of study medication, assessed up to approximately 56 weeks
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Treatment Period: LOU064 25 mg b.i.d.: Patients initially randomized to Remibrutinib (Up to Week 24)
- Double-blind Treatment Period: Placebo: Patients initially randomized to Placebo during the Double-Blind treatment period (Up to Week 24)
- Transitioned to LOU064 25 mg b.i.d.: Patients initially randomized to placebo during the Double-blind treatment period and switched to Remibrutinib during the Open-label treatment period (Weeks 25-52)
Arm/Group | Double-blind Treatment Period: LOU064 25 mg b.i.d. | Double-blind Treatment Period: Placebo | LOU064 25 mg b.i.d. | Transitioned to LOU064 25 mg b.i.d.
Number analyzed (Participants) | 297 | 153 | 297 | 129
Participants
  Patients with at least one Adverse Event (AE) | 205 | 112 | 228 | 71
  Patients with serious or other significant events - Death | 0 | 0 | 0 | 0
  Patients with serious or other significant events - Non-fatal SAE(s) | 10 | 6 | 12 | 2
  Patients with serious or other significant events - Discontinued study treatment due to any AE(s) | 6 | 6 | 13 | 2
  Patients with serious or other significant events - Discontinued study treatment due to any SAE(s) | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study medication up to 28 days after last dose of study medication, assessed up to approximately 56 weeks
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Arm/Group | LOU064 25 mg b.i.d. | Placebo | Transitioned to LOU064 25 mg b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/297 | 0/153 | 0/129
Serious Adverse Events (participants affected / at risk) | 12/297 | 6/153 | 2/129
Other Adverse Events (participants affected / at risk) | 157/297 | 66/153 | 40/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25 mg b.i.d. (N=297) | Placebo (N=153) | Transitioned to LOU064 25 mg b.i.d. (N=129)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LOU064 25 mg b.i.d. (N=297) | Placebo (N=153) | Transitioned to LOU064 25 mg b.i.d. (N=129)
COVID-19 (Infections and infestations) | 62 | 21 | 13
Influenza (Infections and infestations) | 8 | 2 | 4
Nasopharyngitis (Infections and infestations) | 33 | 9 | 3
Sinusitis (Infections and infestations) | 5 | 6 | 1
Suspected COVID-19 (Infections and infestations) | 16 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 22 | 4 | 8
Urinary tract infection (Infections and infestations) | 11 | 4 | 3
Lipase increased (Investigations) | 9 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 4 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 0
Headache (Nervous system disorders) | 22 | 8 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 13 | 0 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT05032157/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT05032157/SAP_001.pdf